CLINICAL TRIAL: NCT06014710
Title: Modelling of Pharyngeal Laryngeal Effectiveness to Assess Swallowing Disorders
Brief Title: Modelling of Pharyngeal Laryngeal Effectiveness
Acronym: Eph-L
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: National Research Agency, France (Other); Institut de Recherche en Informatique de Toulouse (IRIT) (Unknown); Laboratoire parole et langage (Unknown); Swallis Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/22/0091; 2023-A00054-41 (Other: ID-RCB)
Record Dates: First submitted 2023-04-11; First posted 2023-08-28 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Swallowing Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Patients with swallowing disorders and healthy volunteers
  Interventions: Other: Swallowing evaluation

INTERVENTIONS:
Other: Swallowing evaluation — For patients with swallowing disorders: assessment of the swallowing performed according to the available reference examination (videofluoroscopy or nasofibroscopy). In parallel, they will carry the following sensors: microphone, accelerometer, surface electromyography, nasal cannula and pulse oximeter. The subjects will also perform a cough and phonation test and questionnaires. Each subject (or his caregiver) will be contacted by phone once a month for 6 months to monitor the occurrence of complications. The end of study visit at 6 months will be done either at the hospital with a new examination of the swallowing, by telephone, as medically indicated.
  For healthy volunteers: Only one visit is planned for the evaluation of the swallowing with the examination of nasofibroscopy and the installation of the sensors. The procedures (tests, examinations and questionnaires) will be identical to the data collection of the initial visit of patients with swallowing disorders)

SUMMARY:
The purpose of this study is to collect the signals of pharyngeal laryngeal activity through five non-invasive sensors (microphone, accelerometer, surface electromyography (EMG), nasal cannula and oximeter) in order to identify indicators of functional efficiency of swallowing, protection of the lower airways and phonation.

440 patients (subjects with swallowing disorders), spread over 4 centers and 80 healthy subjects spread over 2 centers will be recruited for the study in an interventional research study involving the prospective, multicentric and longitudinal.

Pharyngolaryngeal effectiveness will be measured from 6 indicators identified by examinations or reference tests grouped into 3 functions:

* swallowing: pharyngeal transport capacity (Yale Residue) and Penetration Aspiration Scale (PAS) rated by videofluoroscopy of swallowing (VFS) or flexible endoscopic evaluation of swallowing (FEES);
* airway protection: cough trigger (citric acid test) and cough power (peak expiratory flow);
* phonation: vocal efficiency (maximum phonation time) and velar efficiency (nasal scores).

The signals obtained from the 5 sensors will be annotated. Stochastic modelling based on hidden Markov models will be used initially and followed by the implementation of deep neural networks to model indicators. For the complication's prediction algorithm, deep neural networks will also be used to evaluate signal-based methods.

The expected benefits are to obtain automated recognition of pharyngeal-laryngeal effectiveness to diagnose swallowing disorders using objective and quantifiable indicators, non-invasive devices, to assess the severity of these disorders and to identify the risk of complications.

DETAILED DESCRIPTION:
The process of swallowing is complex and difficult to assess because of its dynamic nature, the lack of specialists and the technical means necessary for its exploration. Thus, the majority of patients with swallowing disorders do not benefit from any specific instrumental evaluation yet essential to the diagnosis of different types of disorders. The precise analysis of the deficit and its causes makes it possible to guide the choice of adaptation or rehabilitation strategies, with the aim of preventing the risk of complications, mainly nutritional (malnutrition) and respiratory (pneumonia). The development of new, more accessible diagnostic techniques would improve access to care for this population. The purpose of this study is to collect the signals of pharyngeal laryngeal activity through five non-invasive sensors (microphone, accelerometer, surface EMG, nasal cannula and oximeter) in order to identify indicators of functional efficiency of swallowing, protection of the lower airways and phonation. Modelling the mechanisms of pharyngeal-laryngeal efficacy through the use of artificial intelligence would provide an automated assessment of disorders and prognostic risk of complications.

Primary objective: From the signals of 5 non-invasive sensors, model a multidimensional scale of pharyngeal-laryngeal efficiency measuring the 3 main functions of pharyngeal-larynx: swallowing function (evaluated by pharyngeal transport and closure of the larynx) ; airway protection function (evaluated by cough reflex and cough power); phonation function (evaluated by voice and velar efficiency)

Secondary Objectives:

* Develop a diagnostic model of different physiopathological mechanisms of swallowing
* Determine an algorithm that can predict the severity of these disorders based on pharyngeal efficacy indicators
* Determine an algorithm capable of predicting the risk of complications from swallowing disorders, based on modelling pharyngeal effectiveness (primary objective) and clinical data

Study design: An interventional research study involving the prospective, multicentric and longitudinal human person to develop a scale of pharyngeal-laryngeal effectiveness measured from signals from 5 non-invasive sensors. The signals will be collected from each participant using the sensors (microphone, accelerometer, nasal cannula, surface EMG and oximeter). Algorithms will be developed from these signals to predict different indicators of pharyngeal-laryngeal efficiency measured by baseline tests. The study population will include patients with swallowing disorders (to identify pathological signal patterns) and healthy volunteers (to identify non-pathological physiological patterns of swallowing mechanisms).

440 patients (subjects with swallowing disorders), spread over 4 centers and 80 healthy subjects spread over 2 centers will be recruited for the study.

Research procedures

For patients with swallowing disorders:

During a hospital visit as part of their care pathway, patients with the criteria will be offered to participate in the research protocol. The subjects who have given their written consent will then carry out their assessment of the swallowing performed according to the available reference examination (videofluoroscopy or nasofibroscopy). In parallel, they will carry the following sensors: microphone, accelerometer, surface electromyography, nasal cannula and pulse oximeter. For research purposes, the subjects will also perform a cough and phonation test and questionnaires. Other data used are collected as part of routine care.

At the end of the assessment, the patient will receive management advice based on the reference exams and his medical record.

Each subject (or his caregiver) will be contacted by phone once a month for 6 months to monitor the occurrence of complications, The end of study visit at 6 months will be done either at the hospital with a new examination of the swallowing, by telephone, as medically indicated.

For healthy volunteers:

Only one visit is planned for the evaluation of the swallowing with the examination of nasofibroscopy and the installation of the sensors. The procedures (tests, examinations and questionnaires) will be identical to the data collection of the initial visit of patients with swallowing disorders)

Duration of the research: The first patient will be included from 2023. The inclusion period is 18 months. Patients will be monitored for 6 months (+/- 2 months) after inclusion Healthy volunteers will have one visit (estimated time: 2H) The total duration of the clinical study is expected to be 26 months

Data analysis: The characteristics of the subjects as well as the various clinical indicators of swallowing and their evolution during monitoring will be described. Development and validation algorithms to model the various pharyngo-laryngeal effectiveness indicators and predictive algorithms of swallowing disorders will be produced using statistical approaches and also using machine learning. The signals obtained from the 5 sensors will be annotated. The signals will be standardized and synchronized to allow the modelling of the sequences corresponding to the following events: swallowing of food, saliva, cough, throat clearing, speech, wet voice. Stochastic modelling based on hidden Markov models will be used initially and followed by the implementation of deep neural networks to model indicators. For the complication's prediction algorithm, deep neural networks will also be used to evaluate signal-based methods.

ELIGIBILITY:
Inclusion criteria for patients with swallowing disorders :

* Indication to perform a swallowing test (suspected or proven swallowing disorder or presence of a complication)
* Able to follow up by phone for 6 months or have a caregiver who can answer for them
* Affiliated subject or beneficiary of the social security system
* Consent to participate obtained in writing and signed by the subject or, if applicable, the next of kin/support person

Inclusion criteria for healthy volunteers :

* No swallowing disorder or discomfort (DHI score<8)
* Affiliated subject or beneficiary of the social security system
* Signed Consent to Participate

Non-inclusion criteria for patients with swallowing disorders :

* Skin lesion(s) at the neck
* Tracheotomy or tracheostomy (laryngectomy)
* Nasogastric probe
* Iodine allergy
* Asthma
* Refusal or any pathology incompatible with passing one of the two reference exams or the sensors used
* Any serious pathology (severe health or behavioral disorders) where, according to the investigator, this could expose participants to additional risks
* Legal protection (guardianship, curators, safeguarding of justice)
* Pregnant and lactating women

Non-inclusion criteria for healthy volunteers :

* Medical history may result in chronic (history of oral-rhino-laryngeal cancer or neurological disease) or temporary (upper respiratory tract infections) swallowing impairment
* Presence of swallowing disorder or discomfort (Deglutition Handicap Index score superior or equal to 8)
* Skin lesion(s) at the neck
* Tracheotomy or tracheostomy (laryngectomy)
* Nasogastric probe
* Iodine allergy
* Asthma
* Refusal or any pathology incompatible with passing one of the two reference exams or the sensors used
* Any serious pathology (severe health or behavioral disorders) where, according to the investigator, this could expose participants to additional risks
* Legal protection (guardianship, curators, safeguarding of justice)
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Swallowing efficacy | Baseline
  Swallowing efficacy : pharyngeal transport capacity (assessed by the Yale Pharyngeal residue severity rating scale). The Yale Pharyngeal residue severity rating scale (YPRSRS) is a 5-point scale ranging from I (none) to V (severe).
Swallowing safety | Baseline
  Swallowing Safety : the Penetration Aspiration Scale (PAS) rated by VFS (videofluoroscopy of swallowing) or FEES (flexible endoscopic evaluation of swallowing). The Penetration Aspiration Scale (PAS) is a 8-point scale ranging from 1 to 8 : 1 is considered the best and 8 the worst
Lung defense reflex | Baseline
  Cough trigger reviewed by citric acid test
Power of cough | Baseline
  Cough power rated by peak expiratory flow in litres per minute
Voice efficiency | Baseline
  Vocal efficiency evaluated by maximum phonation time on the letter "a" held in seconds
Velar efficiency | Baseline
  velar efficiency evaluated by assessment of the sentences without nasal phonemes and sentences with nasal phonemes

SECONDARY OUTCOMES:
Self-assessment of severity of swallowing disorders | Baseline
  Severity of swallowing disorders measured by patient self-assessment with visual analogic scale ranging from 1 = no severity to 10 = very severe.
Severity of swallowing disorders assessed by oropharyngeal swallowing effectiveness scale | Baseline
  Severity of swallowing disorders measured by oropharyngeal swallowing effectiveness scale from baseline studies (FEES or VFS). The OroPharyngeal Swallowing Efficiency (OPSE) is a subjective evaluation of the severity expressed as a percentage of the bolus actually passing through the esophagus according to the formula:
  100% (of the bolus introduced into the mouth) - X% of the bolus having gone astray - Y% of the bolus stagnating in the form of residue
General quality of life assessment | Baseline and 6 months
  Quality of life assessed by euroqol 5-dimension 5-level questionnaire (EQ-5D-5L). The EQ-5D-5L is questionnaire with 5 items from 1 to 5 : 1 is considered the best and 5 the worst and a scale from 100 " the best health you can imagine " to 0 " the worst health you can imagine ".
Quality of life assessment for patients with cancer | Baseline and 6 months
  Quality of life assessed by Cancer Quality of life questionnaire (CLQ-C30) for patients with cancer. The CLQ-C30 questionnaire is composed of 30 items.

CONTACTS AND LOCATIONS:
Overall Officials: Virginie WOISARD, MD, Principal Investigator — University Hospital of Toulouse
Locations (4):
- France (4):
  - University hospital of Bordeaux, Bordeaux
  - University hospital of Rouen, Rouen
  - University Hospital of Toulouse, Toulouse
  - University hospital of Tours, Tours

IPD SHARING:
Plan to Share IPD: No